CLINICAL TRIAL: NCT04927312
Title: A PHASE 3, MULTICENTER, OPEN-LABEL, SINGLE-ARM STUDY TO ASSESS THE EFFICACY AND SAFETY OF CEFTAZIDIME-AVIBACTAM (PF-06947386) PLUS METRONIDAZOLE IN JAPANESE ADULT PATIENTS WITH COMPLICATED INTRA-ABDOMINAL INFECTION REQUIRING HOSPITALIZATION
Brief Title: Study to Assess Efficacy and Safety of PF-06947386 in Japanese Adult Patients With Complicated Intra-abdominal Infection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C3591036
Record Dates: First submitted 2021-06-04; First posted 2021-06-15 (Actual); Results first posted 2024-03-08 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Complicated Intra-abdominal Infection
Keywords: Ceftazidime-avibactam,; Metronidazole,; complicated intra-abdominal infection
MeSH Terms: interventions — Metronidazole

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- PF-06947386 + Metronidazole (Experimental): Multiple intravenous infusion of ceftazidime-avibactam followed by intravenous infusion of metronidazole, repeated every 8 hours for 5-14 days.
  Interventions: Drug: PF-06947386; Drug: Metronidazole

INTERVENTIONS:
Drug: PF-06947386 — Ceftazidime-Avibactam powder for concentrate for solution for infusion 2.0 g/ 0.5 g. Dosage will be adjusted based on renal function after enrollment.
Drug: Metronidazole — Metronidazole 0.5 g solution for injection.

SUMMARY:
Study C3591036 is a Phase 3 study to assess the efficacy and safety of PF-06947386 in Japanese adult patients with complicated intra-abdominal infection requiring hospitalization. This is a multicenter, open-label, single-arm study. All eligible participants will receive intravenous infusion of PF-06947386 followed by intravenous infusion of metronidazole.

ELIGIBILITY:
Inclusion Criteria:

* Participant who is capable of giving signed, dated and timed informed consent (or by their legally acceptable representative)
* Participant aged 20 years or older
* Participant who is willing and able to comply with all scheduled visits, treatment plan, laboratory tests, and other study procedures
* Confirmation of infection by surgical intervention within 24 hours of entry: evidence of systemic inflammatory response; physical findings consistent with intra-abdominal infection; supportive radiologic imaging findings of intra-abdominal infections
* Intraoperative/postoperative enrollment with visual confirmation (presence of pus within the abdominal cavity) of an intra-abdominal infection associated with peritonitis

Exclusion Criteria:

* Participant will undergo surgery for traumatic bowel perforation within 12 hours or perforation of gastroduodenal ulcers within 24 hours. Other intra-abdominal processes that are not infectious.
* Participant has abdominal wall abscess or bowel obstruction without perforation or ischemic bowel without perforation
* Participant whose surgery will include staged abdominal repair, or "open abdomen" technique, or marsupialization.
* Participant has evidence of sepsis with shock not responding to IV fluid challenge or anticipated to require the administration of vasopressors for >24 hours
* Participant has suspected intra-abdominal infections due to fungus, parasites (eg, amebic liver abscess), virus, or tuberculosis
* Participant is considered unlikely to survive the 6- to 8-week study period or has a rapidly progressive or terminal illness
* Participant is pregnant or breastfeeding.
* Participant has received systemic antibacterial agents within the 72-hour period prior to study entry except for cases specified in the protocol such that participant is considered to have failed the previous treatment regimen, or participant has received systemic antibiotic agents no more than 24 hours (no more than one daily dose) within the 72-hour period prior to study entry, etc.
* Estimated CrCL ≤50 mL/min calculated by Cockcroft-Gault method.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-09-15 (Actual); Study Completion 2022-09-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (29):
- Japan (29):
  - Nagoya Ekisaikai Hospital, Nagoya, Aichi-ken
  - National Hospital Organization Nagoya Medical Center, Nagoya, Aichi-ken
  - National Hospital Organization Toyohashi Medical Center, Toyohashi, Aichi-ken
  - Fukuoka Tokushukai Hospital, Kasuga, Fukuoka
  - St.Mary's Hospital, Kurume, Fukuoka
  - Gunma Saiseikai Maebashi Hospital, Maebashi, Gunma
  - Saiseikai Maebashi Hospital, Maebashi, Gunma
  - Teine Keijinkai Hospital, Sapporo, Hokkaido
  - Tsuchiura Kyodo General Hospital, Tsuchiura, Ibaraki
  - Tsuchiura Kyodo General Hospital, Tsuchiura-shi, Ibaraki
  - National Hospital Organization Kanazawa Medical Center, Kanazawa, Ishikawa-ken
  - Kawasaki Saiwai Hospital, Kawasaki-shi, Kanagawa
  - Sagamihara Kyodo Hospital, Sagamihara, Kanagawa
  - National Hospital Organization Yokohama Medical Center, Yokohama, Kanagawa
  - Suwa Red Cross Hospital, Suwa, Nagano
  - National Hospital Organization Nagasaki Medical Center, Ōmura, Nagasaki
  - Nagaoka Chuo General Hospital, Nagaoka, Niigata
  - Naha City Hospital, Naha, Okinawa
  - Rinku General Medical Center, Izumisano, Osaka
  - National Hospital Organization Osaka Minami Medical Center, Kawachi-Nagano, Osaka
  - Yamanashi Prefectural Central Hospital, Kofu, Yamanashi
  - National Hospital Organization Chiba Medical Center, Chiba
  - Fukuoka Wajiro Hospital, Fukuoka
  - National Hospital Organization Kumamoto Medical Center, Kumamoto
  - National Hospital Organization Kyoto Medical Center, Kyoto
  - Okayama City General Medical Center Okayama City Hospital, Okayama
  - Osaka Saiseikai Nakatsu Hospital, Osaka
  - Toyama University Hospital, Toyama
  - Yamagata City Hospital Saiseikan, Yamagata

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Mikamo H, Nakazuru Y, Tabuchi R, Suzuki M, Nagashima M, Tawadrous M, Wible M, Ohta M. Efficacy and safety of ceftazidime-avibactam in combination with metronidazole in Japanese patients with complicated intra-abdominal infection: A phase 3, multicentre, open-label study. J Infect Chemother. 2025 Mar;31(3):102598. doi: 10.1016/j.jiac.2024.102598. Epub 2024 Dec 21. PMID 39710167
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C3591036

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 60 Japanese hospitalized participants with complicated intra-abdominal infection (cIAI) were enrolled in this study.
Groups:
- PF-06947386 + Metronidazole: Participants received intravenous (IV) infusion of PF-06947386 (2.0 gram (g) of ceftazidime and 0.5 g of avibactam) every 8 hours, immediately followed by an IV administration of metronidazole (0.5 g) for 60 minutes. Participants received a minimum of 5 full days (15 doses) of IV study intervention up to a maximum of 14 full days (42 doses) of study intervention.
Period: Overall Study
Arm/Group | PF-06947386 + Metronidazole
Started | 60
Completed | 56
Not Completed | 4
Not completed — Adverse Event | 1
Not completed — Death | 1
Not completed — Withdrawal by Subject | 1
Not completed — Other | 1

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants who received any amount of IV study intervention.
Arm/Group | PF-06947386 + Metronidazole
Number analyzed (Participants) | 60
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.5 (17.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 34
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 60
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 60
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Clinical Response at Test of Cure (TOC) Visit: Clinically Evaluable (CE) Analysis Set
Description: Clinical response: Clinical response of cure was defined as complete resolution or significant improvement of signs and symptoms of the index infection such that no further antimicrobial therapy, drainage, or surgical intervention was necessary. TOC was after 28 calendar days from the day of the first IV infusion, allowed visit window was 28 to 35 calendar days after the day of the first IV infusion; clinical failure: Death related to intra-abdominal infection, Persisting or recurrent infection within the abdomen, Postsurgical wound infections, participant who received treatment with additional antibiotics for ongoing symptoms of intra-abdominal infection; Indeterminate: Study data was not available for evaluation of efficacy for any reason. TOC was after 28 calendar days from the day of the first IV infusion, allowed visit window was 28 to 35 calendar days after the day of the first IV infusion.
Time Frame: TOC: Any day from Day 28 to Day 35
Population: CE analysis set included participants who had an appropriate diagnosis of cIAI; either received therapy for greater than or equal to (>=) 48 hours, with >=80 percent (%) of the scheduled drug administered over number of days administered or received therapy less than (<) 48 hours before discontinuing treatment due to an adverse event (AE).
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06947386 + Metronidazole
Number analyzed (Participants) | 40
Participants
  Clinical Cure | 36
  Clinical Failure | 4
  Indeterminate | 0

2. Secondary Outcome: Percentage of Participants With Clinical Response at End of Treatment (EOT) and Late Follow-up (LFU) Visits: CE Analysis Set
Description: Clinical response: Clinical response of cure was defined as complete resolution or significant improvement of signs and symptoms of the index infection such that no further antimicrobial therapy, drainage, or surgical intervention was necessary. TOC was after 28 calendar days from the day of the first IV infusion, allowed visit window was 28 to 35 calendar days after the day of the first IV infusion; clinical failure: Death related to intra-abdominal infection, Persisting or recurrent infection within the abdomen, Postsurgical wound infections, participant who received treatment with additional antibiotics for ongoing symptoms of intra-abdominal infection; Indeterminate: Study data was not available for evaluation of efficacy for any reason. EOT: within 24 hours after completion of last IV infusion. LFU: after 42 calendar days from the day of the first IV infusion, the allowed visit window was 42 to 49 calendar days from the day of the first IV infusion.
Time Frame: EOT: 24 hours after last IV infusion; LFU: Any day from Day 42 to Day 49
Population: CE analysis set evaluated. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure. Here, "Number Analyzed" signifies participants included in CE analysis set at EOT and LFU respectively.
Measure: Number; unit: Percentage of participants
Arm/Group | PF-06947386 + Metronidazole
Number analyzed (Participants) | 42
Percentage of participants
  EOT, Clinical Cure | 90.5
  EOT, Clinical Failure | 9.5
  EOT, Indeterminate | 0
  LFU, Clinical Cure: number analyzed (Participants) | 40
  LFU, Clinical Cure | 90.0
  LFU, Clinical Failure: number analyzed (Participants) | 40
  LFU, Clinical Failure | 10.0
  LFU, Indeterminate: number analyzed (Participants) | 40
  LFU, Indeterminate | 0

3. Secondary Outcome: Number of Participants With Clinical Response at EOT and LFU Visits: Modified Intent-to-Treat (MITT) Analysis Set
Description: as for outcome 2
Time Frame: EOT: 24 hours after last IV infusion; LFU: Any day from Day 42 to Day 49
Population: MITT analysis set included all enrolled participants who had clinical evidence of cIAI and received any amount of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06947386 + Metronidazole
Number analyzed (Participants) | 59
Participants
  EOT, Clinical Cure | 54
  EOT, Clinical Failure | 4
  EOT, Indeterminate | 1
  LFU, Clinical Cure | 52
  LFU, Clinical Failure | 4
  LFU, Indeterminate | 3

4. Secondary Outcome: Number of Participants With Clinical Response at EOT and LFU Visits: Microbiological Modified Intent-to-Treat (mMITT) Analysis Set
Description: as for outcome 2
Time Frame: EOT: 24 hours after last IV infusion; LFU: Any day from Day 42 to Day 49
Population: mMITT analysis set included all enrolled participant who met the disease definition of cIAI; received any amount of study drug and had at least 1 etiologic pathogen identified at study entry (regardless of isolate susceptibilities).
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06947386 + Metronidazole
Number analyzed (Participants) | 42
Participants
  EOT, Clinical Cure | 38
  EOT, Clinical Failure | 4
  EOT, Indeterminate | 0
  LFU, Clinical Cure | 36
  LFU, Clinical Failure | 4
  LFU, Indeterminate | 2

5. Secondary Outcome: Percentage of Participants With Clinical Response at EOT and LFU Visits: Microbiologically Evaluable (ME) Analysis Set
Description: Clinical response: Clinical response of cure was defined as complete resolution or significant improvement of signs and symptoms of the index infection such that no further antimicrobial therapy, drainage, or surgical intervention was necessary. TOC was after 28 calendar days from the day of the first IV infusion, allowed visit window was 28 to 35 calendar days after the day of the first IV infusion; clinical failure: Death related to intra-abdominal infection, Persisting or recurrent infection within the abdomen, Postsurgical wound infections, participant who received treatment with additional antibiotics for ongoing symptoms of intra-abdominal infection; Indeterminate: Study data was not available for evaluation of efficacy for any reason. LFU: after 42 calendar days from the day of the first IV infusion, the allowed visit window was 42 to 49 calendar days from the day of the first IV infusion.
Time Frame: EOT: 24 hours after last IV infusion; LFU: Any day from Day 42 to Day 49
Population: ME analysis set included participants who were included in a subset of CE participants and had at least 1 Gram-negative aerobic pathogen in the initial/prestudy culture that was susceptible. Here, "Number Analyzed" signifies participants included in ME analysis set at EOT and LFU respectively.
Measure: Number; unit: Percentage of Participants
Arm/Group | PF-06947386 + Metronidazole
Number analyzed (Participants) | 36
Percentage of Participants
  EOT, Clinical Cure | 94.4
  EOT, Clinical Failure | 5.6
  EOT, Indeterminate | 0
  LFU, Clinical Cure: number analyzed (Participants) | 35
  LFU, Clinical Cure | 94.3
  LFU, Clinical Failure: number analyzed (Participants) | 35
  LFU, Clinical Failure | 5.7
  LFU, Indeterminate: number analyzed (Participants) | 35
  LFU, Indeterminate | 0

6. Secondary Outcome: Percentage of Participants With Clinical Response EOT and LFU Visits: Extended Microbiologically Evaluable (eME) Analysis Set
Description: as for outcome 2
Time Frame: EOT: 24 hours after last IV infusion; LFU: Any day from Day 42 to Day 49
Population: eME analysis set included participants who were included in a subset of CE participants and had at least 1 Gram-negative aerobic pathogen in the initial/prestudy culture that is susceptible. Here, "Number Analyzed" signifies participants included in eME analysis set at EOT and LFU respectively.
Measure: Number; unit: Percentage of Participants
Arm/Group | PF-06947386 + Metronidazole
Number analyzed (Participants) | 37
Percentage of Participants
  EOT, Clinical Cure | 94.6
  EOT, Clinical Failure | 5.4
  EOT, Indeterminate | 0
  LFU, Clinical Cure: number analyzed (Participants) | 36
  LFU, Clinical Cure | 94.4
  LFU, Clinical Failure: number analyzed (Participants) | 36
  LFU, Clinical Failure | 5.6
  LFU, Indeterminate: number analyzed (Participants) | 36
  LFU, Indeterminate | 0

7. Secondary Outcome: Number of Participants With Microbiological Response EOT, TOC and LFU Visits: mMITT Analysis Set
Description: Microbiological response: Favorable microbiological response assessments include "eradication", "presumed eradication" and "colonization". Unfavorable microbiological response assessments include "persistence", "persistence with increasing MIC", and "presumed persistence. Indeterminate: Study data are not available for evaluation of efficacy. "Indeterminate" were not included in the denominator. EOT: within 24 hours after completion of last IV infusion. LFU: after 42 calendar days from the day of the first IV infusion, the allowed visit window was 42 to 49 calendar days from the day of the first IV infusion. TOC: after 28 calendar days from the day of the first IV infusion, allowed visit window was 28 to 35 calendar days after the day of the first IV infusion.
Time Frame: EOT: 24 hours after last IV infusion; TOC: Any day from Day 28 to 35; LFU: Any day from Day 42 to Day 49
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06947386 + Metronidazole
Number analyzed (Participants) | 42
Participants
  EOT, Favorable | 38
  EOT, Unfavorable | 4
  EOT, Indeterminate | 0
  TOC, Favorable | 36
  TOC, Unfavorable | 4
  TOC, Indeterminate | 2
  LFU, Favorable | 36
  LFU, Unfavorable | 4
  LFU, Indeterminate | 2

8. Secondary Outcome: Percentage of Participants With Microbiological Response EOT, TOC and LFU Visits: ME Analysis Set
Description: Microbiological response: Favorable microbiological response assessments include "eradication", "presumed eradication" and "colonization". Unfavorable microbiological response assessments include "persistence", "persistence with increasing MIC", and "presumed persistence. Indeterminate: Study data was not available for evaluation of efficacy. "Indeterminate" were not included in the denominator. EOT: within 24 hours after completion of last IV infusion. LFU: after 42 calendar days from the day of the first IV infusion, the allowed visit window was 42 to 49 calendar days from the day of the first IV infusion. TOC: after 28 calendar days from the day of the first IV infusion, allowed visit window was 28 to 35 calendar days after the day of the first IV infusion.
Time Frame: EOT: 24 hours after last IV infusion; TOC: Any day from Day 28 to 35; LFU: Any day from Day 42 to Day 49
Population: ME analysis set included participants who were included in a subset of CE participants and had at least 1 Gram-negative aerobic pathogen in the initial/prestudy culture that was susceptible. Here, "Number Analyzed" signifies participants included in ME analysis set at EOT, TOC and LFU respectively.
Measure: Number; unit: Percentage of Participants
Arm/Group | PF-06947386 + Metronidazole
Number analyzed (Participants) | 36
Percentage of Participants
  EOT, Favorable | 94.4
  EOT, Unfavorable | 5.6
  EOT, Indeterminate | 0
  TOC, Favorable: number analyzed (Participants) | 35
  TOC, Favorable | 94.3
  TOC, Unfavorable: number analyzed (Participants) | 35
  TOC, Unfavorable | 5.7
  TOC, Indeterminate: number analyzed (Participants) | 35
  TOC, Indeterminate | 0
  LFU, Favorable: number analyzed (Participants) | 35
  LFU, Favorable | 94.3
  LFU, Unfavorable: number analyzed (Participants) | 35
  LFU, Unfavorable | 5.7
  LFU, Indeterminate: number analyzed (Participants) | 35
  LFU, Indeterminate | 0

9. Secondary Outcome: Percentage of Participants With Microbiological Response EOT, TOC and LFU Visits: eME Analysis Set
Description: as for outcome 8
Time Frame: EOT: 24 hours after last IV infusion; TOC: Any day from Day 28 to 35; LFU: Any day from Day 42 to Day 49
Population: eME analysis set included participants who were included in a subset of CE participants and had at least 1 Gram-negative aerobic pathogen in the initial/prestudy culture that is susceptible. Here, "Number Analyzed" signifies participants included in eME analysis set at EOT, TOC and LFU respectively.
Measure: Number; unit: Percentage of Participants
Arm/Group | PF-06947386 + Metronidazole
Number analyzed (Participants) | 37
Percentage of Participants
  EOT, Favorable | 94.6
  EOT, Unfavorable | 5.4
  EOT, Indeterminate | 0
  TOC, Favorable: number analyzed (Participants) | 36
  TOC, Favorable | 94.4
  TOC, Unfavorable: number analyzed (Participants) | 36
  TOC, Unfavorable | 5.6
  TOC, Indeterminate: number analyzed (Participants) | 36
  TOC, Indeterminate | 0
  LFU, Favorable: number analyzed (Participants) | 36
  LFU, Favorable | 94.4
  LFU, Unfavorable: number analyzed (Participants) | 36
  LFU, Unfavorable | 5.6
  LFU, Indeterminate: number analyzed (Participants) | 36
  LFU, Indeterminate | 0

10. Secondary Outcome: Percentage of Participants With Favorable Per-Pathogen Microbiological Response at EOT, TOC and LFU Visits: mMITT Analysis Set
Description: Microbiological response: Favorable microbiological response assessments include "eradication", "presumed eradication" and "colonization". Unfavorable microbiological response assessments include "persistence", "persistence with increasing MIC", and "presumed persistence. Indeterminate: Study data was not available for evaluation of efficacy. "Indeterminate" were not included in the denominator. EOT: within 24 hours after completion of last IV infusion. Response of baseline pathogens cultured from intra-abdominal site or blood. A participant can have more than 1 pathogen. LFU: after 42 calendar days from the day of the first IV infusion, the allowed visit window was 42 to 49 calendar days from the day of the first IV infusion. TOC: after 28 calendar days from the day of the first IV infusion, allowed visit window was 28 to 35 calendar days after the day of the first IV infusion.
Time Frame: EOT: 24 hours after last IV infusion; TOC: Any day from Day 28 to 35; LFU: Any day from Day 42 to Day 49
Population: mMITT analysis set:all enrolled participant who met disease definition of cIAI; received any amount of study drug; had at least 1 etiologic pathogen identified at study entry."Overall Number of Participants Analyzed": participants evaluable for this outcome measure however all participants reported under 'Overall Number of Participants Analyzed' contributed data to table but may not have evaluable data for every row. "Number Analyzed":participants included in eME analysis set at EOT, TOC & LFU.
Measure: Number; unit: Percentage of Participants
Arm/Group | PF-06947386 + Metronidazole
Number analyzed (Participants) | 42
Percentage of Participants
  EOT, Enterobacter Aerogenes: number analyzed (Participants) | 2
  EOT, Enterobacter Aerogenes | 100.0
  EOT, Escherichia Coli: number analyzed (Participants) | 31
  EOT, Escherichia Coli | 93.5
  EOT, Klebsiella Oxytoca: number analyzed (Participants) | 1
  EOT, Klebsiella Oxytoca | 100.0
  EOT, Klebsiella Pneumoniae: number analyzed (Participants) | 5
  EOT, Klebsiella Pneumoniae | 100.0
  EOT, Proteus Mirabilis: number analyzed (Participants) | 1
  EOT, Proteus Mirabilis | 100.0
  EOT, Proteus Penneri: number analyzed (Participants) | 1
  EOT, Proteus Penneri | 100.0
  EOT, Proteus Vulgaris: number analyzed (Participants) | 1
  EOT, Proteus Vulgaris | 100.0
  EOT, Raoultella Planticola: number analyzed (Participants) | 2
  EOT, Raoultella Planticola | 50.0
  EOT, Pseudomonas Aeruginosa: number analyzed (Participants) | 6
  EOT, Pseudomonas Aeruginosa | 100.0
  TOC, Enterobacter Aerogenes: number analyzed (Participants) | 2
  TOC, Enterobacter Aerogenes | 100.0
  TOC, Escherichia Coli: number analyzed (Participants) | 30
  TOC, Escherichia Coli | 93.3
  TOC, Klebsiella Oxytoca: number analyzed (Participants) | 1
  TOC, Klebsiella Oxytoca | 100.0
  TOC, Klebsiella Pneumoniae: number analyzed (Participants) | 5
  TOC, Klebsiella Pneumoniae | 100.0
  TOC, Proteus Mirabilis: number analyzed (Participants) | 1
  TOC, Proteus Mirabilis | 100.0
  TOC, Proteus Penneri: number analyzed (Participants) | 1
  TOC, Proteus Penneri | 100.0
  TOC, Proteus Vulgaris: number analyzed (Participants) | 1
  TOC, Proteus Vulgaris | 100.0
  TOC, Raoultella Planticola: number analyzed (Participants) | 1
  TOC, Raoultella Planticola | 0.0
  TOC, Pseudomonas Aeruginosa: number analyzed (Participants) | 6
  TOC, Pseudomonas Aeruginosa | 100.0
  LFU, Enterobacter Aerogenes: number analyzed (Participants) | 2
  LFU, Enterobacter Aerogenes | 100.0
  LFU, Escherichia Coli: number analyzed (Participants) | 30
  LFU, Escherichia Coli | 93.3
  LFU, Klebsiella Oxytoca: number analyzed (Participants) | 1
  LFU, Klebsiella Oxytoca | 100.0
  LFU, Klebsiella Pneumoniae: number analyzed (Participants) | 5
  LFU, Klebsiella Pneumoniae | 100.0
  LFU, Proteus Mirabilis: number analyzed (Participants) | 1
  LFU, Proteus Mirabilis | 100.0
  LFU, Proteus Penneri: number analyzed (Participants) | 1
  LFU, Proteus Penneri | 100.0
  LFU, Proteus Vulgaris: number analyzed (Participants) | 1
  LFU, Proteus Vulgaris | 100.0
  LFU, Raoultella Planticola: number analyzed (Participants) | 1
  LFU, Raoultella Planticola | 0.0
  LFU, Pseudomonas Aeruginosa: number analyzed (Participants) | 6
  LFU, Pseudomonas Aeruginosa | 100.0

11. Secondary Outcome: Percentage of Participants With Favorable Per-Pathogen Microbiological Response at EOT, TOC and LFU Visits: ME Analysis Set
Description: Microbiological response: Favorable microbiological response assessments include "eradication", "presumed eradication" and "colonization". Unfavorable microbiological response assessments include "persistence", "persistence with increasing MIC", and "presumed persistence. Indeterminate: Study data are not available for evaluation of efficacy. "Indeterminate" were not included in the denominator. EOT: within 24 hours after completion of last IV infusion. Response of baseline pathogens cultured from intra-abdominal site or blood. A participant can have more than 1 pathogen. LFU: after 42 calendar days from the day of the first IV infusion, the allowed visit window was 42 to 49 calendar days from the day of the first IV infusion. TOC: after 28 calendar days from the day of the first IV infusion, allowed visit window was 28 to 35 calendar days after the day of the first IV infusion.
Time Frame: EOT: 24 hours after last IV infusion; TOC: Any day from Day 28 to 35; LFU: Any day from Day 42 to Day 49
Population: ME analysis set: participants who were included in subset of CE participants & had at least 1 Gram-negative aerobic pathogen in the initial/prestudy culture that was susceptible. "Overall Number of Participants Analyzed":participants evaluable for this outcome measure however all participants reported under 'Overall Number of Participants Analyzed' contributed data to table but may not have evaluable data for every row. "Number Analyzed":participants included in ME analysis set at EOT,TOC & LFU
Measure: Number; unit: Percentage of Participants
Arm/Group | PF-06947386 + Metronidazole
Number analyzed (Participants) | 36
Percentage of Participants
  EOT, Enterobacter Aerogenes: number analyzed (Participants) | 2
  EOT, Enterobacter Aerogenes | 100.0
  EOT, Escherichia Coli: number analyzed (Participants) | 31
  EOT, Escherichia Coli | 93.5
  EOT, Klebsiella Oxytoca: number analyzed (Participants) | 1
  EOT, Klebsiella Oxytoca | 100.0
  EOT, Klebsiella Pneumoniae: number analyzed (Participants) | 5
  EOT, Klebsiella Pneumoniae | 100.0
  EOT, Proteus Mirabilis: number analyzed (Participants) | 1
  EOT, Proteus Mirabilis | 100.0
  EOT, Proteus Penneri: number analyzed (Participants) | 1
  EOT, Proteus Penneri | 100.0
  EOT, Proteus Vulgaris: number analyzed (Participants) | 1
  EOT, Proteus Vulgaris | 100.0
  EOT, Raoultella Planticola: number analyzed (Participants) | 2
  EOT, Raoultella Planticola | 50.0
  EOT, Pseudomonas Aeruginosa: number analyzed (Participants) | 6
  EOT, Pseudomonas Aeruginosa | 100.0
  TOC, Enterobacter Aerogenes: number analyzed (Participants) | 2
  TOC, Enterobacter Aerogenes | 100.0
  TOC, Escherichia Coli: number analyzed (Participants) | 30
  TOC, Escherichia Coli | 93.3
  TOC, Klebsiella Oxytoca: number analyzed (Participants) | 1
  TOC, Klebsiella Oxytoca | 100.0
  TOC, Klebsiella Pneumoniae: number analyzed (Participants) | 5
  TOC, Klebsiella Pneumoniae | 100.0
  TOC, Proteus Mirabilis: number analyzed (Participants) | 1
  TOC, Proteus Mirabilis | 100.0
  TOC, Proteus Penneri: number analyzed (Participants) | 1
  TOC, Proteus Penneri | 100.0
  TOC, Proteus Vulgaris: number analyzed (Participants) | 1
  TOC, Proteus Vulgaris | 100.0
  TOC, Raoultella Planticola: number analyzed (Participants) | 1
  TOC, Raoultella Planticola | 0.0
  TOC, Pseudomonas Aeruginosa: number analyzed (Participants) | 6
  TOC, Pseudomonas Aeruginosa | 100.0
  LFU, Enterobacter Aerogenes: number analyzed (Participants) | 2
  LFU, Enterobacter Aerogenes | 100.0
  LFU, Escherichia Coli: number analyzed (Participants) | 30
  LFU, Escherichia Coli | 93.3
  LFU, Klebsiella Oxytoca: number analyzed (Participants) | 1
  LFU, Klebsiella Oxytoca | 100.0
  LFU, Klebsiella Pneumoniae: number analyzed (Participants) | 5
  LFU, Klebsiella Pneumoniae | 100.0
  LFU, Proteus Mirabilis: number analyzed (Participants) | 1
  LFU, Proteus Mirabilis | 100.0
  LFU, Proteus Penneri: number analyzed (Participants) | 1
  LFU, Proteus Penneri | 100.0
  LFU, Proteus Vulgaris: number analyzed (Participants) | 1
  LFU, Proteus Vulgaris | 100.0
  LFU, Raoultella Planticola: number analyzed (Participants) | 1
  LFU, Raoultella Planticola | 0.0
  LFU, Pseudomonas Aeruginosa: number analyzed (Participants) | 6
  LFU, Pseudomonas Aeruginosa | 100.0

12. Secondary Outcome: Percentage of Participants With Favorable Per-Pathogen Microbiological Response at EOT, TOC and LFU Visits: eME Analysis Set
Description: as for outcome 10
Time Frame: EOT: 24 hours after last IV infusion; TOC: Any day from Day 28 to 35; LFU: Any day from Day 42 to Day 49
Population: eME analysis set: participants who were included in subset of CE participants & had at least 1 Gram-negative aerobic pathogen in initial/prestudy culture that is susceptible. Overall Number of Participants Analyzed":participants evaluable for this outcome measure however all participants reported under 'Overall Number of Participants Analyzed' contributed data to table but may not have evaluable data for every row. "Number Analyzed": participants included in eME analysis set at EOT, TOC & LFU.
Measure: Number; unit: Percentage of Participants
Arm/Group | PF-06947386 + Metronidazole
Number analyzed (Participants) | 37
Percentage of Participants
  EOT, Enterobacter Aerogenes: number analyzed (Participants) | 2
  EOT, Enterobacter Aerogenes | 100.0
  EOT, Escherichia Coli: number analyzed (Participants) | 31
  EOT, Escherichia Coli | 93.5
  EOT, Klebsiella Oxytoca: number analyzed (Participants) | 1
  EOT, Klebsiella Oxytoca | 100.0
  EOT, Klebsiella Pneumoniae: number analyzed (Participants) | 5
  EOT, Klebsiella Pneumoniae | 100.0
  EOT, Proteus Mirabilis: number analyzed (Participants) | 1
  EOT, Proteus Mirabilis | 100.0
  EOT, Proteus Penneri: number analyzed (Participants) | 1
  EOT, Proteus Penneri | 100.0
  EOT, Proteus Vulgaris: number analyzed (Participants) | 1
  EOT, Proteus Vulgaris | 100.0
  EOT, Raoultella Planticola: number analyzed (Participants) | 2
  EOT, Raoultella Planticola | 50.0
  EOT, Pseudomonas Aeruginosa: number analyzed (Participants) | 6
  EOT, Pseudomonas Aeruginosa | 100.0
  TOC, Enterobacter Aerogenes: number analyzed (Participants) | 2
  TOC, Enterobacter Aerogenes | 100.0
  TOC, Escherichia Coli: number analyzed (Participants) | 30
  TOC, Escherichia Coli | 93.3
  TOC, Klebsiella Oxytoca: number analyzed (Participants) | 1
  TOC, Klebsiella Oxytoca | 100.0
  TOC, Klebsiella Pneumoniae: number analyzed (Participants) | 5
  TOC, Klebsiella Pneumoniae | 100.0
  TOC, Proteus Mirabilis: number analyzed (Participants) | 1
  TOC, Proteus Mirabilis | 100.0
  TOC, Proteus Penneri: number analyzed (Participants) | 1
  TOC, Proteus Penneri | 100.0
  TOC, Proteus Vulgaris: number analyzed (Participants) | 1
  TOC, Proteus Vulgaris | 100.0
  TOC, Raoultella Planticola: number analyzed (Participants) | 1
  TOC, Raoultella Planticola | 0.0
  TOC, Pseudomonas Aeruginosa: number analyzed (Participants) | 6
  TOC, Pseudomonas Aeruginosa | 100.0
  LFU, Enterobacter Aerogenes: number analyzed (Participants) | 2
  LFU, Enterobacter Aerogenes | 100.0
  LFU, Escherichia Coli: number analyzed (Participants) | 30
  LFU, Escherichia Coli | 93.3
  LFU, Klebsiella Oxytoca: number analyzed (Participants) | 1
  LFU, Klebsiella Oxytoca | 100.0
  LFU, Klebsiella Pneumoniae: number analyzed (Participants) | 5
  LFU, Klebsiella Pneumoniae | 100.0
  LFU, Proteus Mirabilis: number analyzed (Participants) | 1
  LFU, Proteus Mirabilis | 100.0
  LFU, Proteus Penneri: number analyzed (Participants) | 1
  LFU, Proteus Penneri | 100.0
  LFU, Proteus Vulgaris: number analyzed (Participants) | 1
  LFU, Proteus Vulgaris | 100.0
  LFU, Raoultella Planticola: number analyzed (Participants) | 1
  LFU, Raoultella Planticola | 0.0
  LFU, Pseudomonas Aeruginosa: number analyzed (Participants) | 6
  LFU, Pseudomonas Aeruginosa | 100.0

13. Secondary Outcome: Percentage of Participants With Favorable Per-Pathogen Microbiological Response by Minimum Inhibitory Concentration (MIC) Categories at EOT, TOC and LFU Visits: mMITT Analysis Set
Description: as for outcome 8
Time Frame: EOT: 24 hours after last IV infusion; TOC: Any day from Day 28 to 35; LFU: Any day from Day 42 to Day 49
Population: as for outcome 10
Measure: Number; unit: Percentage of Participants
Arm/Group | PF-06947386 + Metronidazole
Number analyzed (Participants) | 42
Percentage of Participants
  EOT, Enterobacter Aerogenes, Susceptible: number analyzed (Participants) | 2
  EOT, Enterobacter Aerogenes, Susceptible | 100.0
  EOT, Enterobacter Aerogenes, Intermediate: number analyzed (Participants) | 0
  EOT, Enterobacter Aerogenes, Resistant: number analyzed (Participants) | 0
  EOT, Escherichia Coli, Susceptible: number analyzed (Participants) | 30
  EOT, Escherichia Coli, Susceptible | 93.3
  EOT, Escherichia Coli, Intermediate: number analyzed (Participants) | 0
  EOT, Escherichia Coli, Resistant: number analyzed (Participants) | 0
  EOT, Klebsiella Oxytoca, Susceptible: number analyzed (Participants) | 1
  EOT, Klebsiella Oxytoca, Susceptible | 100.0
  EOT, Klebsiella Oxytoca, Intermediate: number analyzed (Participants) | 0
  EOT, Klebsiella Oxytoca, Resistant: number analyzed (Participants) | 0
  EOT, Klebsiella Pneumoniae, Susceptible: number analyzed (Participants) | 5
  EOT, Klebsiella Pneumoniae, Susceptible | 100.0
  EOT, Klebsiella Pneumoniae, Intermediate: number analyzed (Participants) | 0
  EOT, Klebsiella Pneumoniae, Resistant: number analyzed (Participants) | 0
  EOT, Proteus Mirabilis, Susceptible: number analyzed (Participants) | 1
  EOT, Proteus Mirabilis, Susceptible | 100.0
  EOT, Proteus Mirabilis, Intermediate: number analyzed (Participants) | 0
  EOT, Proteus Mirabilis, Resistant: number analyzed (Participants) | 0
  EOT, Proteus Penneri, Susceptible: number analyzed (Participants) | 1
  EOT, Proteus Penneri, Susceptible | 100.0
  EOT, Proteus Penneri, Intermediate: number analyzed (Participants) | 0
  EOT, Proteus Penneri, Resistant: number analyzed (Participants) | 0
  EOT, Proteus Vulgaris, Susceptible: number analyzed (Participants) | 1
  EOT, Proteus Vulgaris, Susceptible | 100.0
  EOT, Proteus Vulgaris, Intermediate: number analyzed (Participants) | 0
  EOT, Proteus Vulgaris, Resistant: number analyzed (Participants) | 0
  EOT, Raoultella Planticola, Susceptible: number analyzed (Participants) | 2
  EOT, Raoultella Planticola, Susceptible | 50.0
  EOT, Raoultella Planticola, Intermediate: number analyzed (Participants) | 0
  EOT, Raoultella Planticola, Resistant: number analyzed (Participants) | 0
  EOT, Pseudomonas Aeruginosa, Susceptible: number analyzed (Participants) | 6
  EOT, Pseudomonas Aeruginosa, Susceptible | 100.0
  EOT, Pseudomonas Aeruginosa, Intermediate: number analyzed (Participants) | 0
  EOT, Pseudomonas Aeruginosa, Resistant: number analyzed (Participants) | 0
  TOC, Enterobacter Aerogenes, Susceptible: number analyzed (Participants) | 2
  TOC, Enterobacter Aerogenes, Susceptible | 100.0
  TOC, Enterobacter Aerogenes, Intermediate: number analyzed (Participants) | 0
  TOC, Enterobacter Aerogenes, Resistant: number analyzed (Participants) | 0
  TOC, Escherichia Coli, Susceptible: number analyzed (Participants) | 29
  TOC, Escherichia Coli, Susceptible | 93.1
  TOC, Escherichia Coli, Intermediate: number analyzed (Participants) | 0
  TOC, Escherichia Coli, Resistant: number analyzed (Participants) | 0
  TOC, Klebsiella Oxytoca, Susceptible: number analyzed (Participants) | 1
  TOC, Klebsiella Oxytoca, Susceptible | 100.0
  TOC, Klebsiella Oxytoca, Intermediate: number analyzed (Participants) | 0
  TOC, Klebsiella Oxytoca, Resistant: number analyzed (Participants) | 0
  TOC, Klebsiella Pneumoniae, Susceptible: number analyzed (Participants) | 5
  TOC, Klebsiella Pneumoniae, Susceptible | 100.0
  TOC, Klebsiella Pneumoniae, Intermediate: number analyzed (Participants) | 0
  TOC, Klebsiella Pneumoniae, Resistant: number analyzed (Participants) | 0
  TOC, Proteus Mirabilis, Susceptible: number analyzed (Participants) | 1
  TOC, Proteus Mirabilis, Susceptible | 100.0
  TOC, Proteus Mirabilis, Intermediate: number analyzed (Participants) | 0
  TOC, Proteus Mirabilis, Resistant: number analyzed (Participants) | 0
  TOC, Proteus Penneri, Susceptible: number analyzed (Participants) | 1
  TOC, Proteus Penneri, Susceptible | 100.0
  TOC, Proteus Penneri, Intermediate: number analyzed (Participants) | 0
  TOC, Proteus Penneri, Resistant: number analyzed (Participants) | 0
  TOC, Proteus Vulgaris, Susceptible: number analyzed (Participants) | 1
  TOC, Proteus Vulgaris, Susceptible | 100.0
  TOC, Proteus Vulgaris, Intermediate: number analyzed (Participants) | 0
  TOC, Proteus Vulgaris, Resistant: number analyzed (Participants) | 0
  TOC, Raoultella Planticola, Susceptible: number analyzed (Participants) | 1
  TOC, Raoultella Planticola, Susceptible | 0.0
  TOC, Raoultella Planticola, Intermediate: number analyzed (Participants) | 0
  TOC, Raoultella Planticola, Resistant: number analyzed (Participants) | 0
  TOC, Pseudomonas Aeruginosa, Susceptible: number analyzed (Participants) | 6
  TOC, Pseudomonas Aeruginosa, Susceptible | 100.0
  TOC, Pseudomonas Aeruginosa, Intermediate: number analyzed (Participants) | 0
  TOC, Pseudomonas Aeruginosa, Resistant: number analyzed (Participants) | 0
  LFU, Enterobacter Aerogenes, Susceptible: number analyzed (Participants) | 2
  LFU, Enterobacter Aerogenes, Susceptible | 100.0
  LFU, Enterobacter Aerogenes, Intermediate: number analyzed (Participants) | 0
  LFU, Enterobacter Aerogenes, Resistant: number analyzed (Participants) | 0
  LFU, Escherichia Coli, Susceptible: number analyzed (Participants) | 29
  LFU, Escherichia Coli, Susceptible | 93.1
  LFU, Escherichia Coli, Intermediate: number analyzed (Participants) | 0
  LFU, Escherichia Coli, Resistant: number analyzed (Participants) | 0
  LFU, Klebsiella Oxytoca, Susceptible: number analyzed (Participants) | 1
  LFU, Klebsiella Oxytoca, Susceptible | 100.0
  LFU, Klebsiella Oxytoca, Intermediate: number analyzed (Participants) | 0
  LFU, Klebsiella Oxytoca, Resistant: number analyzed (Participants) | 0
  LFU, Klebsiella Pneumoniae, Susceptible: number analyzed (Participants) | 5
  LFU, Klebsiella Pneumoniae, Susceptible | 100.0
  LFU, Klebsiella Pneumoniae, Intermediate: number analyzed (Participants) | 0
  LFU, Klebsiella Pneumoniae, Resistant: number analyzed (Participants) | 0
  LFU, Proteus Mirabilis, Susceptible: number analyzed (Participants) | 1
  LFU, Proteus Mirabilis, Susceptible | 100.0
  LFU, Proteus Mirabilis, Intermediate: number analyzed (Participants) | 0
  LFU, Proteus Mirabilis, Resistant: number analyzed (Participants) | 0
  LFU, Proteus Penneri, Susceptible: number analyzed (Participants) | 1
  LFU, Proteus Penneri, Susceptible | 100.0
  LFU, Proteus Penneri, Intermediate: number analyzed (Participants) | 0
  LFU, Proteus Penneri, Resistant: number analyzed (Participants) | 0
  LFU, Proteus Vulgaris, Susceptible: number analyzed (Participants) | 1
  LFU, Proteus Vulgaris, Susceptible | 100.0
  LFU, Proteus Vulgaris, Intermediate: number analyzed (Participants) | 0
  LFU, Proteus Vulgaris, Resistant: number analyzed (Participants) | 0
  LFU, Raoultella Planticola, Susceptible: number analyzed (Participants) | 1
  LFU, Raoultella Planticola, Susceptible | 0.0
  LFU, Raoultella Planticola, Intermediate: number analyzed (Participants) | 0
  LFU, Raoultella Planticola, Resistant: number analyzed (Participants) | 0
  LFU, Pseudomonas Aeruginosa, Susceptible: number analyzed (Participants) | 6
  LFU, Pseudomonas Aeruginosa, Susceptible | 100.0
  LFU, Pseudomonas Aeruginosa, Intermediate: number analyzed (Participants) | 0
  LFU, Pseudomonas Aeruginosa, Resistant: number analyzed (Participants) | 0

14. Secondary Outcome: Percentage of Participants With Favorable Per-Pathogen Microbiological Response by MIC Categories at EOT, TOC and LFU Visits: ME Analysis Set
Description: as for outcome 8
Time Frame: EOT: 24 hours after last IV infusion; TOC: Any day from Day 28 to 35; LFU: Any day from Day 42 to Day 49
Population: as for outcome 11
Measure: Number; unit: Percentage of Participants
Arm/Group | PF-06947386 + Metronidazole
Number analyzed (Participants) | 36
Percentage of Participants
  EOT, Enterobacter Aerogenes, Susceptible: number analyzed (Participants) | 2
  EOT, Enterobacter Aerogenes, Susceptible | 100.0
  EOT, Enterobacter Aerogenes, Intermediate: number analyzed (Participants) | 0
  EOT, Enterobacter Aerogenes, Resistant: number analyzed (Participants) | 0
  EOT, Escherichia Coli, Susceptible: number analyzed (Participants) | 30
  EOT, Escherichia Coli, Susceptible | 93.3
  EOT, Escherichia Coli, Intermediate: number analyzed (Participants) | 0
  EOT, Escherichia Coli, Resistant: number analyzed (Participants) | 0
  EOT, Klebsiella Oxytoca, Susceptible: number analyzed (Participants) | 1
  EOT, Klebsiella Oxytoca, Susceptible | 100.0
  EOT, Klebsiella Oxytoca, Intermediate: number analyzed (Participants) | 0
  EOT, Klebsiella Oxytoca, Resistant: number analyzed (Participants) | 0
  EOT, Klebsiella Pneumoniae, Susceptible: number analyzed (Participants) | 5
  EOT, Klebsiella Pneumoniae, Susceptible | 100.0
  EOT, Klebsiella Pneumoniae, Intermediate: number analyzed (Participants) | 0
  EOT, Klebsiella Pneumoniae, Resistant: number analyzed (Participants) | 0
  EOT, Proteus Mirabilis, Susceptible: number analyzed (Participants) | 1
  EOT, Proteus Mirabilis, Susceptible | 100.0
  EOT, Proteus Mirabilis, Intermediate: number analyzed (Participants) | 0
  EOT, Proteus Mirabilis, Resistant: number analyzed (Participants) | 0
  EOT, Proteus Penneri, Susceptible: number analyzed (Participants) | 1
  EOT, Proteus Penneri, Susceptible | 100.0
  EOT, Proteus Penneri, Intermediate: number analyzed (Participants) | 0
  EOT, Proteus Penneri, Resistant: number analyzed (Participants) | 0
  EOT, Proteus Vulgaris, Susceptible: number analyzed (Participants) | 1
  EOT, Proteus Vulgaris, Susceptible | 100.0
  EOT, Proteus Vulgaris, Intermediate: number analyzed (Participants) | 0
  EOT, Proteus Vulgaris, Resistant: number analyzed (Participants) | 0
  EOT, Raoultella Planticola, Susceptible: number analyzed (Participants) | 2
  EOT, Raoultella Planticola, Susceptible | 50.0
  EOT, Raoultella Planticola, Intermediate: number analyzed (Participants) | 0
  EOT, Raoultella Planticola, Resistant: number analyzed (Participants) | 0
  EOT, Pseudomonas Aeruginosa, Susceptible: number analyzed (Participants) | 6
  EOT, Pseudomonas Aeruginosa, Susceptible | 100.0
  EOT, Pseudomonas Aeruginosa, Intermediate: number analyzed (Participants) | 0
  EOT, Pseudomonas Aeruginosa, Resistant: number analyzed (Participants) | 0
  TOC, Enterobacter Aerogenes, Susceptible: number analyzed (Participants) | 2
  TOC, Enterobacter Aerogenes, Susceptible | 100.0
  TOC, Enterobacter Aerogenes, Intermediate: number analyzed (Participants) | 0
  TOC, Enterobacter Aerogenes, Resistant: number analyzed (Participants) | 0
  TOC, Escherichia Coli, Susceptible: number analyzed (Participants) | 29
  TOC, Escherichia Coli, Susceptible | 93.1
  TOC, Escherichia Coli, Intermediate: number analyzed (Participants) | 0
  TOC, Escherichia Coli, Resistant: number analyzed (Participants) | 0
  TOC, Klebsiella Oxytoca, Susceptible: number analyzed (Participants) | 1
  TOC, Klebsiella Oxytoca, Susceptible | 100.0
  TOC, Klebsiella Oxytoca, Intermediate: number analyzed (Participants) | 0
  TOC, Klebsiella Oxytoca, Resistant: number analyzed (Participants) | 0
  TOC, Klebsiella Pneumoniae, Susceptible: number analyzed (Participants) | 5
  TOC, Klebsiella Pneumoniae, Susceptible | 100.0
  TOC, Klebsiella Pneumoniae, Intermediate: number analyzed (Participants) | 0
  TOC, Klebsiella Pneumoniae, Resistant: number analyzed (Participants) | 0
  TOC, Proteus Mirabilis, Susceptible: number analyzed (Participants) | 1
  TOC, Proteus Mirabilis, Susceptible | 100.0
  TOC, Proteus Mirabilis, Intermediate: number analyzed (Participants) | 0
  TOC, Proteus Mirabilis, Resistant: number analyzed (Participants) | 0
  TOC, Proteus Penneri, Susceptible: number analyzed (Participants) | 1
  TOC, Proteus Penneri, Susceptible | 100.0
  TOC, Proteus Penneri, Intermediate: number analyzed (Participants) | 0
  TOC, Proteus Penneri, Resistant: number analyzed (Participants) | 0
  TOC, Proteus Vulgaris, Susceptible: number analyzed (Participants) | 1
  TOC, Proteus Vulgaris, Susceptible | 100.0
  TOC, Proteus Vulgaris, Intermediate: number analyzed (Participants) | 0
  TOC, Proteus Vulgaris, Resistant: number analyzed (Participants) | 0
  TOC, Raoultella Planticola, Susceptible: number analyzed (Participants) | 1
  TOC, Raoultella Planticola, Susceptible | 0.0
  TOC, Raoultella Planticola, Intermediate: number analyzed (Participants) | 0
  TOC, Raoultella Planticola, Resistant: number analyzed (Participants) | 0
  TOC, Pseudomonas Aeruginosa, Susceptible: number analyzed (Participants) | 6
  TOC, Pseudomonas Aeruginosa, Susceptible | 100.0
  TOC, Pseudomonas Aeruginosa, Intermediate: number analyzed (Participants) | 0
  TOC, Pseudomonas Aeruginosa, Resistant: number analyzed (Participants) | 0
  LFU, Enterobacter Aerogenes, Susceptible: number analyzed (Participants) | 2
  LFU, Enterobacter Aerogenes, Susceptible | 100.0
  LFU, Enterobacter Aerogenes, Intermediate: number analyzed (Participants) | 0
  LFU, Enterobacter Aerogenes, Resistant: number analyzed (Participants) | 0
  LFU, Escherichia Coli, Susceptible: number analyzed (Participants) | 29
  LFU, Escherichia Coli, Susceptible | 93.1
  LFU, Escherichia Coli, Intermediate: number analyzed (Participants) | 0
  LFU, Escherichia Coli, Resistant: number analyzed (Participants) | 0
  LFU, Klebsiella Oxytoca, Susceptible: number analyzed (Participants) | 1
  LFU, Klebsiella Oxytoca, Susceptible | 100.0
  LFU, Klebsiella Oxytoca, Intermediate: number analyzed (Participants) | 0
  LFU, Klebsiella Oxytoca, Resistant: number analyzed (Participants) | 0
  LFU, Klebsiella Pneumoniae, Susceptible: number analyzed (Participants) | 5
  LFU, Klebsiella Pneumoniae, Susceptible | 100.0
  LFU, Klebsiella Pneumoniae, Intermediate: number analyzed (Participants) | 0
  LFU, Klebsiella Pneumoniae, Resistant: number analyzed (Participants) | 0
  LFU, Proteus Mirabilis, Susceptible: number analyzed (Participants) | 1
  LFU, Proteus Mirabilis, Susceptible | 100.0
  LFU, Proteus Mirabilis, Intermediate: number analyzed (Participants) | 0
  LFU, Proteus Mirabilis, Resistant: number analyzed (Participants) | 0
  LFU, Proteus Penneri, Susceptible: number analyzed (Participants) | 1
  LFU, Proteus Penneri, Susceptible | 100.0
  LFU, Proteus Penneri, Intermediate: number analyzed (Participants) | 0
  LFU, Proteus Penneri, Resistant: number analyzed (Participants) | 0
  LFU, Proteus Vulgaris, Susceptible: number analyzed (Participants) | 1
  LFU, Proteus Vulgaris, Susceptible | 100.0
  LFU, Proteus Vulgaris, Intermediate: number analyzed (Participants) | 0
  LFU, Proteus Vulgaris, Resistant: number analyzed (Participants) | 0
  LFU, Raoultella Planticola, Susceptible: number analyzed (Participants) | 1
  LFU, Raoultella Planticola, Susceptible | 0.0
  LFU, Raoultella Planticola, Intermediate: number analyzed (Participants) | 0
  LFU, Raoultella Planticola, Resistant: number analyzed (Participants) | 0
  LFU, Pseudomonas Aeruginosa, Susceptible: number analyzed (Participants) | 6
  LFU, Pseudomonas Aeruginosa, Susceptible | 100.0
  LFU, Pseudomonas Aeruginosa, Intermediate: number analyzed (Participants) | 0
  LFU, Pseudomonas Aeruginosa, Resistant: number analyzed (Participants) | 0

15. Secondary Outcome: Percentage of Participants With Favorable Per-Pathogen Microbiological Response by MIC Categories at EOT, TOC and LFU Visits: eME Analysis Set
Description: as for outcome 8
Time Frame: EOT: 24 hours after last IV infusion; TOC: Any day from Day 28 to 35; LFU: Any day from Day 42 to Day 49
Population: as for outcome 12
Measure: Number; unit: Percentage of Participants
Arm/Group | PF-06947386 + Metronidazole
Number analyzed (Participants) | 37
Percentage of Participants
  EOT, Enterobacter Aerogenes, Susceptible: number analyzed (Participants) | 2
  EOT, Enterobacter Aerogenes, Susceptible | 100.0
  EOT, Enterobacter Aerogenes, Intermediate: number analyzed (Participants) | 0
  EOT, Enterobacter Aerogenes, Resistant: number analyzed (Participants) | 0
  EOT, Escherichia Coli, Susceptible: number analyzed (Participants) | 30
  EOT, Escherichia Coli, Susceptible | 93.3
  EOT, Escherichia Coli, Intermediate: number analyzed (Participants) | 0
  EOT, Escherichia Coli, Resistant: number analyzed (Participants) | 0
  EOT, Klebsiella Oxytoca, Susceptible: number analyzed (Participants) | 1
  EOT, Klebsiella Oxytoca, Susceptible | 100.0
  EOT, Klebsiella Oxytoca, Intermediate: number analyzed (Participants) | 0
  EOT, Klebsiella Oxytoca, Resistant: number analyzed (Participants) | 0
  EOT, Klebsiella Pneumoniae, Susceptible: number analyzed (Participants) | 5
  EOT, Klebsiella Pneumoniae, Susceptible | 100.0
  EOT, Klebsiella Pneumoniae, Intermediate: number analyzed (Participants) | 0
  EOT, Klebsiella Pneumoniae, Resistant: number analyzed (Participants) | 0
  EOT, Proteus Mirabilis, Susceptible: number analyzed (Participants) | 1
  EOT, Proteus Mirabilis, Susceptible | 100.0
  EOT, Proteus Mirabilis, Intermediate: number analyzed (Participants) | 0
  EOT, Proteus Mirabilis, Resistant: number analyzed (Participants) | 0
  EOT, Proteus Penneri, Susceptible: number analyzed (Participants) | 1
  EOT, Proteus Penneri, Susceptible | 100.0
  EOT, Proteus Penneri, Intermediate: number analyzed (Participants) | 0
  EOT, Proteus Penneri, Resistant: number analyzed (Participants) | 0
  EOT, Proteus Vulgaris, Susceptible: number analyzed (Participants) | 1
  EOT, Proteus Vulgaris, Susceptible | 100.0
  EOT, Proteus Vulgaris, Intermediate: number analyzed (Participants) | 0
  EOT, Proteus Vulgaris, Resistant: number analyzed (Participants) | 0
  EOT, Raoultella Planticola, Susceptible: number analyzed (Participants) | 2
  EOT, Raoultella Planticola, Susceptible | 50.0
  EOT, Raoultella Planticola, Intermediate: number analyzed (Participants) | 0
  EOT, Raoultella Planticola, Resistant: number analyzed (Participants) | 0
  EOT, Pseudomonas Aeruginosa, Susceptible: number analyzed (Participants) | 6
  EOT, Pseudomonas Aeruginosa, Susceptible | 100.0
  EOT, Pseudomonas Aeruginosa, Intermediate: number analyzed (Participants) | 0
  EOT, Pseudomonas Aeruginosa, Resistant: number analyzed (Participants) | 0
  TOC, Enterobacter Aerogenes, Susceptible: number analyzed (Participants) | 2
  TOC, Enterobacter Aerogenes, Susceptible | 100.0
  TOC, Enterobacter Aerogenes, Intermediate: number analyzed (Participants) | 0
  TOC, Enterobacter Aerogenes, Resistant: number analyzed (Participants) | 0
  TOC, Escherichia Coli, Susceptible: number analyzed (Participants) | 29
  TOC, Escherichia Coli, Susceptible | 93.1
  TOC, Escherichia Coli, Intermediate: number analyzed (Participants) | 0
  TOC, Escherichia Coli, Resistant: number analyzed (Participants) | 0
  TOC, Klebsiella Oxytoca, Susceptible: number analyzed (Participants) | 1
  TOC, Klebsiella Oxytoca, Susceptible | 100.0
  TOC, Klebsiella Oxytoca, Intermediate: number analyzed (Participants) | 0
  TOC, Klebsiella Oxytoca, Resistant: number analyzed (Participants) | 0
  TOC, Klebsiella Pneumoniae, Susceptible: number analyzed (Participants) | 5
  TOC, Klebsiella Pneumoniae, Susceptible | 100.0
  TOC, Klebsiella Pneumoniae, Intermediate: number analyzed (Participants) | 0
  TOC, Klebsiella Pneumoniae, Resistant: number analyzed (Participants) | 0
  TOC, Proteus Mirabilis, Susceptible: number analyzed (Participants) | 1
  TOC, Proteus Mirabilis, Susceptible | 100.0
  TOC, Proteus Mirabilis, Intermediate: number analyzed (Participants) | 0
  TOC, Proteus Mirabilis, Resistant: number analyzed (Participants) | 0
  TOC, Proteus Penneri, Susceptible: number analyzed (Participants) | 1
  TOC, Proteus Penneri, Susceptible | 100.0
  TOC, Proteus Penneri, Intermediate: number analyzed (Participants) | 0
  TOC, Proteus Penneri, Resistant: number analyzed (Participants) | 0
  TOC, Proteus Vulgaris, Susceptible: number analyzed (Participants) | 1
  TOC, Proteus Vulgaris, Susceptible | 100.0
  TOC, Proteus Vulgaris, Intermediate: number analyzed (Participants) | 0
  TOC, Proteus Vulgaris, Resistant: number analyzed (Participants) | 0
  TOC, Raoultella Planticola, Susceptible: number analyzed (Participants) | 1
  TOC, Raoultella Planticola, Susceptible | 0.0
  TOC, Raoultella Planticola, Intermediate: number analyzed (Participants) | 0
  TOC, Raoultella Planticola, Resistant: number analyzed (Participants) | 0
  TOC, Pseudomonas Aeruginosa, Susceptible: number analyzed (Participants) | 6
  TOC, Pseudomonas Aeruginosa, Susceptible | 100.0
  TOC, Pseudomonas Aeruginosa, Intermediate: number analyzed (Participants) | 0
  TOC, Pseudomonas Aeruginosa, Resistant: number analyzed (Participants) | 0
  LFU, Enterobacter Aerogenes, Susceptible: number analyzed (Participants) | 2
  LFU, Enterobacter Aerogenes, Susceptible | 100.0
  LFU, Enterobacter Aerogenes, Intermediate: number analyzed (Participants) | 0
  LFU, Enterobacter Aerogenes, Resistant: number analyzed (Participants) | 0
  LFU, Escherichia Coli, Susceptible: number analyzed (Participants) | 29
  LFU, Escherichia Coli, Susceptible | 93.1
  LFU, Escherichia Coli, Intermediate: number analyzed (Participants) | 0
  LFU, Escherichia Coli, Resistant: number analyzed (Participants) | 0
  LFU, Klebsiella Oxytoca, Susceptible: number analyzed (Participants) | 1
  LFU, Klebsiella Oxytoca, Susceptible | 100.0
  LFU, Klebsiella Oxytoca, Intermediate: number analyzed (Participants) | 0
  LFU, Klebsiella Oxytoca, Resistant: number analyzed (Participants) | 0
  LFU, Klebsiella Pneumoniae, Susceptible: number analyzed (Participants) | 5
  LFU, Klebsiella Pneumoniae, Susceptible | 100.0
  LFU, Klebsiella Pneumoniae, Intermediate: number analyzed (Participants) | 0
  LFU, Klebsiella Pneumoniae, Resistant: number analyzed (Participants) | 0
  LFU, Proteus Mirabilis, Susceptible: number analyzed (Participants) | 1
  LFU, Proteus Mirabilis, Susceptible | 100.0
  LFU, Proteus Mirabilis, Intermediate: number analyzed (Participants) | 0
  LFU, Proteus Mirabilis, Resistant: number analyzed (Participants) | 0
  LFU, Proteus Penneri, Susceptible: number analyzed (Participants) | 1
  LFU, Proteus Penneri, Susceptible | 100.0
  LFU, Proteus Penneri, Intermediate: number analyzed (Participants) | 0
  LFU, Proteus Penneri, Resistant: number analyzed (Participants) | 0
  LFU, Proteus Vulgaris, Susceptible: number analyzed (Participants) | 1
  LFU, Proteus Vulgaris, Susceptible | 100.0
  LFU, Proteus Vulgaris, Intermediate: number analyzed (Participants) | 0
  LFU, Proteus Vulgaris, Resistant: number analyzed (Participants) | 0
  LFU, Raoultella Planticola, Susceptible: number analyzed (Participants) | 1
  LFU, Raoultella Planticola, Susceptible | 0.0
  LFU, Raoultella Planticola, Intermediate: number analyzed (Participants) | 0
  LFU, Raoultella Planticola, Resistant: number analyzed (Participants) | 0
  LFU, Pseudomonas Aeruginosa, Susceptible: number analyzed (Participants) | 6
  LFU, Pseudomonas Aeruginosa, Susceptible | 100.0
  LFU, Pseudomonas Aeruginosa, Intermediate: number analyzed (Participants) | 0
  LFU, Pseudomonas Aeruginosa, Resistant: number analyzed (Participants) | 0

16. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (AEs) and Serious AEs (SAEs)
Description: An AE was any untoward medical occurrence in a participant or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. SAE was defined as any untoward medical occurrence that, at any dose that resulted in death, was life-threatening, inpatient hospitalization or prolongation of existing hospitalization, persistent disability/incapacity, a congenital anomaly/birth defect as per medical or scientific judgment. AEs included both SAEs and non-SAEs. TEAE was defined as an AE that emerges or worsened during the effective duration of treatment. All events that started on or after the first dosing day were flagged as TEAEs.
Time Frame: Up to Day 49
Population: Safety analysis set included all participants who received any amount of IV study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06947386 + Metronidazole
Number analyzed (Participants) | 60
Participants
  AEs | 42
  SAEs | 3

17. Secondary Outcome: All-cause Mortality
Description: Number of participants with death is presented.
Time Frame: Up to Day 49
Population: Safety analysis set included all participants who received any amount of IV study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06947386 + Metronidazole
Number analyzed (Participants) | 60
Participants | 1

18. Secondary Outcome: Number of Participants Who Discontinued Treatment and Study Due to Adverse Events
Description: Number of participants who discontinued treatment and study due to adverse events is presented.
Time Frame: Up to Day 49
Population: Safety analysis set included all participants who received any amount of IV study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06947386 + Metronidazole
Number analyzed (Participants) | 60
Participants
  Discontinued Treatment due to AE | 0
  Discontinued study due to AE | 2

19. Secondary Outcome: Change From Baseline in Vital Sign Parameters at Day 2 to 14, EOT, TOC and, LFU Visits: Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP)
Description: A semiautomated recording device was used to measure SBP and DBP with participant in a supine position after at least 5 minutes of rest.
Time Frame: Baseline, Day 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, and EOT: 24 hours after last IV infusion; TOC: Any day from Day 28 to 35; LFU: Any day from Day 42 to Day 49
Population: Safety analysis set included all participants who received any amount of IV study intervention. Here, "Number Analyzed" signifies participants included in safety analysis set at EOT, TOC and LFU respectively. Here, "Number Analyzed" signifies number of participants evaluable for specified rows.
Measure: Mean (Standard Deviation); unit: Millimeters of Mercury
Arm/Group | PF-06947386 + Metronidazole
Number analyzed (Participants) | 60
Millimeters of Mercury
  Baseline, SBP | 119.0 (17.73)
  Day 2, SBP | 3.8 (16.05)
  Day 3, SBP: number analyzed (Participants) | 59
  Day 3, SBP | 6.1 (20.44)
  Day 4, SBP: number analyzed (Participants) | 59
  Day 4, SBP | 8.0 (18.27)
  Day 5, SBP: number analyzed (Participants) | 59
  Day 5, SBP | 8.2 (18.26)
  Day 6, SBP: number analyzed (Participants) | 42
  Day 6, SBP | 2.2 (22.92)
  Day 7, SBP: number analyzed (Participants) | 21
  Day 7, SBP | 2.8 (21.61)
  Day 8, SBP: number analyzed (Participants) | 14
  Day 8, SBP | 4.9 (21.14)
  Day 9, SBP: number analyzed (Participants) | 5
  Day 9, SBP | -9.6 (20.61)
  Day 10, SBP: number analyzed (Participants) | 5
  Day 10, SBP | -8.6 (23.86)
  Day 11, SBP: number analyzed (Participants) | 4
  Day 11, SBP | -11.8 (16.50)
  Day 12, SBP: number analyzed (Participants) | 3
  Day 12, SBP | -16.3 (27.57)
  Day 13, SBP: number analyzed (Participants) | 3
  Day 13, SBP | -10.7 (35.50)
  Day 14, SBP: number analyzed (Participants) | 2
  Day 14, SBP | -20.0 (33.94)
  EOT, SBP: number analyzed (Participants) | 59
  EOT, SBP | 2.1 (17.56)
  TOC, SBP: number analyzed (Participants) | 57
  TOC, SBP | 2.1 (19.34)
  LFU, SBP: number analyzed (Participants) | 56
  LFU, SBP | 4.7 (18.78)
  Baseline, DBP | 70.6 (12.90)
  Day 2, DBP | 0.1 (11.31)
  Day 3, DBP: number analyzed (Participants) | 59
  Day 3, DBP | 2.4 (12.77)
  Day 4, DBP: number analyzed (Participants) | 59
  Day 4, DBP | 4.8 (15.13)
  Day 5, DBP: number analyzed (Participants) | 59
  Day 5, DBP | 4.0 (13.90)
  Day 6, DBP: number analyzed (Participants) | 42
  Day 6, DBP | 2.0 (16.36)
  Day 7, DBP: number analyzed (Participants) | 21
  Day 7, DBP | 4.4 (17.53)
  Day 8, DBP: number analyzed (Participants) | 14
  Day 8, DBP | 8.5 (14.90)
  Day 9, DBP: number analyzed (Participants) | 5
  Day 9, DBP | 0.2 (21.05)
  Day 10, DBP: number analyzed (Participants) | 5
  Day 10, DBP | -3.4 (23.10)
  Day 11, DBP: number analyzed (Participants) | 4
  Day 11, DBP | 2.3 (24.80)
  Day 12, DBP: number analyzed (Participants) | 3
  Day 12, DBP | -5.0 (23.30)
  Day 13, DBP: number analyzed (Participants) | 3
  Day 13, DBP | -7.0 (32.19)
  Day 14, DBP: number analyzed (Participants) | 2
  Day 14, DBP | -9.5 (43.13)
  EOT, DBP: number analyzed (Participants) | 59
  EOT, DBP | 0.7 (12.74)
  TOC, DBP: number analyzed (Participants) | 57
  TOC, DBP | 2.9 (13.26)
  LFU, DBP: number analyzed (Participants) | 56
  LFU, DBP | 3.4 (13.86)

20. Secondary Outcome: Change From Baseline in Vital Sign Parameters at Day 2 to 14, EOT, TOC and, LFU Visits: Pulse Rate
Description: Pulse rate was measured for in a supine position preceded by at least 5 minutes of rest for the participant.
Time Frame: as for outcome 19
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | PF-06947386 + Metronidazole
Number analyzed (Participants) | 60
Beats per minute
  Baseline | 82.6 (13.50)
  Day 2 | -4.8 (11.54)
  Day 3: number analyzed (Participants) | 59
  Day 3 | -7.1 (13.04)
  Day 4: number analyzed (Participants) | 59
  Day 4 | -8.9 (14.92)
  Day 5: number analyzed (Participants) | 59
  Day 5 | -11.3 (15.46)
  Day 6: number analyzed (Participants) | 42
  Day 6 | -12.4 (15.61)
  Day 7: number analyzed (Participants) | 21
  Day 7 | -11.0 (18.09)
  Day 8: number analyzed (Participants) | 14
  Day 8 | -9.1 (14.69)
  Day 9: number analyzed (Participants) | 5
  Day 9 | -12.0 (20.25)
  Day 10: number analyzed (Participants) | 5
  Day 10 | -8.0 (29.50)
  Day 11: number analyzed (Participants) | 4
  Day 11 | -12.3 (24.57)
  Day 12: number analyzed (Participants) | 3
  Day 12 | -18.7 (35.36)
  Day 13: number analyzed (Participants) | 3
  Day 13 | -18.0 (37.51)
  Day 14: number analyzed (Participants) | 2
  Day 14 | -24.5 (53.03)
  EOT: number analyzed (Participants) | 59
  EOT | -8.7 (16.56)
  TOC: number analyzed (Participants) | 57
  TOC | -8.8 (16.43)
  LFU: number analyzed (Participants) | 56
  LFU | -9.4 (16.07)

21. Secondary Outcome: Change From Baseline in Vital Sign Parameters at Day 2 to 14, EOT, TOC and, LFU Visits: Weight
Description: Body weight was measured using a balance scale.
Time Frame: as for outcome 19
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: Kilograms
Arm/Group | PF-06947386 + Metronidazole
Number analyzed (Participants) | 60
Kilograms
  Baseline | 62.05 (12.975)
  Day 2: number analyzed (Participants) | 17
  Day 2 | 0.64 (1.587)
  Day 3: number analyzed (Participants) | 11
  Day 3 | 0.68 (1.927)
  Day 4: number analyzed (Participants) | 11
  Day 4 | 0.34 (1.578)
  Day 5: number analyzed (Participants) | 21
  Day 5 | 0.39 (1.949)
  Day 6: number analyzed (Participants) | 12
  Day 6 | 0.82 (1.593)
  Day 7: number analyzed (Participants) | 6
  Day 7 | 1.55 (2.415)
  Day 8: number analyzed (Participants) | 3
  Day 8 | 1.80 (3.894)
  Day 9: number analyzed (Participants) | 1
  Day 9 | 5.80 (NA) — Standard deviation could not be calculated for a single participant.
  Day 10: number analyzed (Participants) | 1
  Day 10 | 5.00 (NA) — Standard deviation could not be calculated for a single participant.
  Day 11: number analyzed (Participants) | 1
  Day 11 | 5.40 (NA) — Standard deviation could not be calculated for a single participant.
  Day 12: number analyzed (Participants) | 2
  Day 12 | -0.05 (5.303)
  Day 13: number analyzed (Participants) | 2
  Day 13 | 1.35 (4.455)
  Day 14: number analyzed (Participants) | 0
  EOT: number analyzed (Participants) | 0
  TOC: number analyzed (Participants) | 0
  LFU: number analyzed (Participants) | 0

22. Secondary Outcome: Change From Baseline in Vital Sign Parameters at Day 2 to 14, EOT, TOC and, LFU Visits: Temperature
Description: Temperature was measured in a supine position, after the participant had rest for at least 5 minutes.
Time Frame: as for outcome 19
Population: Safety analysis set included all participants who received any amount of IV study intervention. Here, "Number Analyzed" signifies participants included in safety analysis set at EOT, TOC and LFU respectively. Here, "Number Analyzed" signifies participants evaluable for specified rows.
Measure: Mean (Standard Deviation); unit: Degree Celsius
Arm/Group | PF-06947386 + Metronidazole
Number analyzed (Participants) | 60
Degree Celsius
  Baseline | 37.01 (0.643)
  Day 2 | 0.33 (0.653)
  Day 3: number analyzed (Participants) | 59
  Day 3 | 0.09 (0.650)
  Day 4: number analyzed (Participants) | 59
  Day 4 | -0.05 (0.679)
  Day 5: number analyzed (Participants) | 59
  Day 5 | -0.12 (0.659)
  Day 6: number analyzed (Participants) | 46
  Day 6 | -0.29 (0.782)
  Day 7: number analyzed (Participants) | 21
  Day 7 | -0.20 (0.846)
  Day 8: number analyzed (Participants) | 15
  Day 8 | -0.19 (0.607)
  Day 9: number analyzed (Participants) | 5
  Day 9 | -0.12 (0.698)
  Day 10: number analyzed (Participants) | 5
  Day 10 | -0.26 (0.811)
  Day 11: number analyzed (Participants) | 4
  Day 11 | -0.30 (0.739)
  Day 12: number analyzed (Participants) | 3
  Day 12 | 0.13 (0.321)
  Day 13: number analyzed (Participants) | 3
  Day 13 | -0.27 (0.493)
  Day 14: number analyzed (Participants) | 2
  Day 14 | -0.10 (0.141)
  EOT: number analyzed (Participants) | 59
  EOT | -0.38 (0.711)
  TOC: number analyzed (Participants) | 57
  TOC | -0.58 (0.766)
  LFU: number analyzed (Participants) | 56
  LFU | -0.54 (0.684)

23. Secondary Outcome: Change From Baseline in Vital Sign Parameters at Day 2 to 14, EOT, TOC and, LFU Visits: Respiratory Rate
Description: Respiratory rate was measured in a supine position, after the participant had rest for at least 5 minutes.
Time Frame: as for outcome 19
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: Breaths per minute
Arm/Group | PF-06947386 + Metronidazole
Number analyzed (Participants) | 60
Breaths per minute
  Baseline | 17.8 (3.39)
  Day 2 | 0.4 (5.91)
  Day 3: number analyzed (Participants) | 59
  Day 3 | -0.4 (4.41)
  Day 4: number analyzed (Participants) | 59
  Day 4 | -1.1 (3.97)
  Day 5: number analyzed (Participants) | 59
  Day 5 | -0.5 (4.79)
  Day 6: number analyzed (Participants) | 42
  Day 6 | -1.3 (3.90)
  Day 7: number analyzed (Participants) | 20
  Day 7 | -1.6 (3.63)
  Day 8: number analyzed (Participants) | 14
  Day 8 | -1.1 (2.66)
  Day 9: number analyzed (Participants) | 5
  Day 9 | -2.8 (3.27)
  Day 10: number analyzed (Participants) | 5
  Day 10 | 0.2 (3.19)
  Day 11: number analyzed (Participants) | 4
  Day 11 | -1.8 (4.19)
  Day 12: number analyzed (Participants) | 3
  Day 12 | -3.3 (4.16)
  Day 13: number analyzed (Participants) | 3
  Day 13 | -0.3 (4.93)
  Day 14: number analyzed (Participants) | 2
  Day 14 | 0.5 (9.19)
  EOT: number analyzed (Participants) | 58
  EOT | -0.6 (4.30)
  TOC: number analyzed (Participants) | 57
  TOC | -1.2 (4.15)
  LFU: number analyzed (Participants) | 56
  LFU | -1.6 (3.88)

24. Secondary Outcome: Number of Participants With Laboratory Test Abnormalities
Description: Criteria for abnormal laboratory values for chemistry parameters: Bilirubin >1.5*upper limit of normal (ULN), direct Bilirubin >1.5*ULN, aspartate aminotransferase, alanine aminotransferase, alkaline phosphatase >3.0*ULN, total protein and albumin <0.8*lower limit of normal (LLN), urea nitrogen and creatinine >1.3*ULN, sodium >0.95*LLN, potassium >0.9*LLN and >1.1*ULN, calcium >0.9*LLN, glucose > 1.5*LLN; hematology parameters: Hemoglobin, hematocrit, erythrocytes <0.8*LLN, platelets <0.5*LLN and > 1.75*ULN, leukocytes <0.6*LLN and <0.6*LLN, lymphocytes <0.8* LLN, lymphocytes/leukocytes <0.8* LLN and >1.2*ULN, neutrophils >1.2*ULN, neutrophils/leukocytes <0.8*LLN and >1.2* ULN, basophils/leukocytes >1.2*ULN, eosinophils >1.2*ULN, eosinophils/leukocytes >1.2*ULN, monocytes and monocytes/leukocytes >1.2*ULN; Criteria for abnormal laboratory values for urinalysis parameters: urine glucose, >=1, urine protein >=1, urine Hemoglobin>=1.
Time Frame: Up to Day 49
Population: Safety analysis set included all participants who received any amount of IV study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06947386 + Metronidazole
Number analyzed (Participants) | 60
Participants | 60

25. Secondary Outcome: Plasma Concentration of Avibactam
Description: Plasma concentrations of avibactam was measured by nominal sampling window.
Time Frame: Day 3, Day 4, and Combination of Day 3 and 4: 15 minutes before or after infusion, 30-90 minutes after infusion, 300-360 minutes after infusion
Population: Pharmacokinetic (PK) analysis set included all participants who have at least 1 plasma concentration data value available for either Ceftazidime or Avibactam. Overall number of participants analyzed signifies participants evaluable for this outcome measure. 'Number Analyzed' signifies participants evaluable for specified rows.
Measure: Mean (Standard Deviation); unit: Nanograms per milliliter
Arm/Group | PF-06947386 + Metronidazole
Number analyzed (Participants) | 58
Nanograms per milliliter
  Day 3, 15 minutes before or after: number analyzed (Participants) | 32
  Day 3, 15 minutes before or after | 13810 (5911.5)
  Day 3, 30-90 minutes after: number analyzed (Participants) | 27
  Day 3, 30-90 minutes after | 8321 (3776.9)
  Day 3, 300-360 minutes after: number analyzed (Participants) | 31
  Day 3, 300-360 minutes after | 1148 (708.04)
  Day 4, 15 minutes before or after: number analyzed (Participants) | 25
  Day 4, 15 minutes before or after | 13940 (4352.1)
  Day 4, 30-90 minutes after: number analyzed (Participants) | 30
  Day 4, 30-90 minutes after | 7897 (2926.5)
  Day 4, 300-360 minutes after: number analyzed (Participants) | 27
  Day 4, 300-360 minutes after | 1651 (2195.6)
  Day 3 and Day 4, 15 minutes before or after: number analyzed (Participants) | 57
  Day 3 and Day 4, 15 minutes before or after | 13870 (5240.9)
  Day 3 and Day 4, 30-90 minutes after: number analyzed (Participants) | 57
  Day 3 and Day 4, 30-90 minutes after | 8098 (3332.2)
  Day 3 and 4, 300-360 minutes after | 1382 (1589.6)

26. Secondary Outcome: Plasma Concentration of Ceftazidime
Description: Plasma concentrations of ceftazidime was measured by nominal sampling window.
Time Frame: as for outcome 25
Population: PK analysis set included all participants who have at least 1 plasma concentration data value available for either Ceftazidime or Avibactam. Overall number of participants analyzed signifies participants evaluable for this outcome measure. Here, "Number Analyzed" signifies participants evaluable for specified rows.
Measure: Mean (Standard Deviation); unit: Nanograms per milliliter
Arm/Group | PF-06947386 + Metronidazole
Number analyzed (Participants) | 58
Nanograms per milliliter
  Day 3, 15 minutes before or after: number analyzed (Participants) | 32
  Day 3, 15 minutes before or after | 72940 (21323)
  Day 3, 30-90 minutes after: number analyzed (Participants) | 27
  Day 3, 30-90 minutes after | 48800 (16611)
  Day 3, 300-360 minutes after: number analyzed (Participants) | 31
  Day 3, 300-360 minutes after | 10030 (5852.5)
  Day 4, 15 minutes before or after: number analyzed (Participants) | 25
  Day 4, 15 minutes before or after | 76680 (26157)
  Day 4, 30-90 minutes after: number analyzed (Participants) | 30
  Day 4, 30-90 minutes after | 49190 (13095)
  Day 4, 300-360 minutes after: number analyzed (Participants) | 27
  Day 4, 300-360 minutes after | 13920 (13135)
  Day 3 and Day 4, 15 minutes before or after: number analyzed (Participants) | 57
  Day 3 and Day 4, 15 minutes before or after | 74580 (23418)
  Day 3 and Day 4, 30-90 minutes after: number analyzed (Participants) | 57
  Day 3 and Day 4, 30-90 minutes after | 49010 (14729)
  Day 3 and Day 4, 300-360 minutes after | 11840 (10028)

27. Other Pre Specified Outcome: Number of Participants With Clinical Response at TOC Visit: MITT Analysis Set
Description: Clinical response: Clinical response of cure was defined as complete resolution or significant improvement of signs and symptoms of the index infection such that no further antimicrobial therapy, drainage, or surgical intervention was necessary. TOC was after 28 calendar days from the day of the first IV infusion, allowed visit window was 28 to 35 calendar days after the day of the first IV infusion; clinical failure: Death related to intra-abdominal infection, Persisting or recurrent infection within the abdomen, Postsurgical wound infections, participant who received treatment with additional antibiotics for ongoing symptoms of intra-abdominal infection; Indeterminate: Study data was not available for evaluation of efficacy for any reason. TOC: after 28 calendar days from the day of the first IV infusion, allowed visit window was 28 to 35 calendar days after the day of the first IV infusion.
Time Frame: TOC: Any day from Day 28 to Day 35
Population: MITT analysis set included all enrolled participants who had clinical evidence of cIAI.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06947386 + Metronidazole
Number analyzed (Participants) | 59
Participants
  TOC, Clinical Cure | 52
  TOC, Clinical Failure | 4
  TOC, Indeterminate | 3

28. Other Pre Specified Outcome: Number of Participants With Clinical Response at TOC Visit: mMITT Analysis Set
Description: as for outcome 27
Time Frame: TOC: Any day from Day 28 to Day 35
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06947386 + Metronidazole
Number analyzed (Participants) | 42
Participants
  TOC, Clinical Cure | 36
  TOC, Clinical Failure | 4
  TOC, Indeterminate | 2

29. Other Pre Specified Outcome: Number of Participants With Clinical Response at TOC: ME Analysis Set
Description: as for outcome 27
Time Frame: TOC: Any day from Day 28 to Day 35
Population: ME analysis set included participants who were included in a subset of CE participants and had at least 1 Gram-negative aerobic pathogen in the initial/prestudy culture that was susceptible.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06947386 + Metronidazole
Number analyzed (Participants) | 35
Participants
  TOC, Clinical Cure | 33
  TOC, Clinical Failure | 2
  TOC, Indeterminate | 0

30. Other Pre Specified Outcome: Number of Participants With Clinical Response at TOC: eME Analysis Set
Description: as for outcome 27
Time Frame: TOC: Any day from Day 28 to Day 35
Population: eME analysis set included participants who were included in a subset of CE participants and had at least 1 Gram-negative aerobic pathogen in the initial/prestudy culture that is susceptible.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06947386 + Metronidazole
Number analyzed (Participants) | 36
Participants
  TOC, Clinical Cure | 34
  TOC, Clinical Failure | 2
  TOC, Indeterminate | 0

31. Other Pre Specified Outcome: Number of Participants With Clinical Response at EOT, TOC and LFU Visits: Sepsis Participants Subset
Description: Clinical response of cure was defined as complete resolution or significant improvement of signs & symptoms of index infection such that no further antimicrobial therapy, drainage, or surgical intervention was necessary. TOC was after 28 calendar days from day of 1st IV infusion, allowed visit window was 28¬-35 calendar days after day of 1st IV infusion; clinical failure: Death related to intra-abdominal infection, Persisting or recurrent infection within abdomen, Postsurgical wound infections, participant who received treatment with additional antibiotics for ongoing symptom of intra-abdominal infection; Indeterminate:Study data was not available for evaluation of efficacy for any reason. EOT: within 24 hours after completion of last IV infusion. LFU:after 42 calendar days from day of 1st IV infusion, allowed visit window was 42-49 calendar days from 1st IV infusion. TOC:after 28 calendar days from 1st IV infusion, allowed visit window was 28-35 calendar days after 1st IV infusion.
Time Frame: EOT: 24 hours after last IV infusion; TOC: Any day from Day 28 to 35; LFU: Any day from Day 42 to Day 49
Population: Sepsis participants subset included participants who satisfied clinical & microbiological criteria; total score >=2 in Sequential Organ Failure Assessment (SOFA) for intensive care unit (ICU) participants, 2 items or more in quick SOFA (qSOFA) for non-ICU participants; most relevant pathogens (aerobic Gram-negative bacteria -either Enterobacterales or aerobic Gram-negative pathogens other than Enterobacterales) isolated from blood at Baseline regardless of susceptibility.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06947386 + Metronidazole
Number analyzed (Participants) | 2
Participants
  EOT, Clinical Cure | 2
  EOT, Clinical Failure | 0
  EOT, Indeterminate | 0
  TOC, Clinical Cure | 2
  TOC, Clinical Failure | 0
  TOC, Indeterminate | 0
  LFU, Clinical Cure | 2
  LFU, Clinical Failure | 0
  LFU, Indeterminate | 0

32. Other Pre Specified Outcome: Number of Participants With Clinical Response at EOT, TOC and LFU Visits: Sepsis Evaluable Participants Subset
Description: as for outcome 31
Time Frame: EOT: 24 hours after last IV infusion; TOC: Any day from Day 28 to 35; LFU: Any day from Day 42 to Day 49
Population: Sepsis evaluable participants subset: participants who satisfied both clinical and microbiological criteria; Clinical: at least one criteria at Baseline. 1) body temperature >=38 degree Celsius or <36 degree Celsius, 2) WBC >12000 cells/mm3 or <4000 cells/mm3, or immature neutrophil >10%, 3) heart rate >90 beats per minute (bpm), 4) SBP <90mmHg, 5) C-reactive protein (CRP) >=20 mg/dL. Microbiological: The most relevant pathogens isolated from blood at Baseline regardless of susceptibility.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06947386 + Metronidazole
Number analyzed (Participants) | 1
Participants
  EOT, Clinical Cure | 1
  EOT, Clinical Failure | 0
  EOT, Indeterminate | 0
  TOC, Clinical Cure | 1
  TOC, Clinical Failure | 0
  TOC, Indeterminate | 0
  LFU, Clinical Cure | 1
  LFU, Clinical Failure | 0
  LFU, Indeterminate | 0

33. Other Pre Specified Outcome: Number of Participants With Microbiological Response EOT, TOC and LFU Visits: Sepsis Participants Subset
Description: Microbiological response: Favorable microbiological response assessments include "eradication", "presumed eradication" and "colonization". Unfavorable microbiological response assessments include "persistence", "persistence with increasing MIC", and "presumed persistence. Indeterminate: Study data are not available for evaluation of efficacy. EOT: within 24 hours after completion of last IV infusion. LFU: after 42 calendar days from the day of the first IV infusion, the allowed visit window was 42 to 49 calendar days from the day of the first IV infusion. TOC: after 28 calendar days from the day of the first IV infusion, allowed visit window was 28 to 35 calendar days after the day of the first IV infusion.
Time Frame: EOT: 24 hours after last IV infusion; TOC: Any day from Day 28 to 35; LFU: Any day from Day 42 to Day 49
Population: Sepsis participants subset included participants who satisfied clinical & microbiological criteria; total score >=2 in SOFA for ICU participants, 2 items or more in qSOFA for non-ICU participants; most relevant pathogens (aerobic Gram-negative bacteria -either Enterobacterales or aerobic Gram-negative pathogens other than Enterobacterales) isolated from blood at Baseline regardless of susceptibility.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06947386 + Metronidazole
Number analyzed (Participants) | 2
Participants
  EOT, Favorable | 2
  EOT, Unfavorable | 0
  EOT, Indeterminate | 0
  TOC, Favorable | 2
  TOC, Unfavorable | 0
  TOC, Indeterminate | 0
  LFU, Favorable | 2
  LFU, Unfavorable | 0
  LFU, Indeterminate | 0

34. Other Pre Specified Outcome: Number of Participants With Microbiological Response EOT, TOC and LFU Visits: Sepsis Evaluable Participants Subset
Description: as for outcome 33
Time Frame: EOT: 24 hours after last IV infusion; TOC: Any day from Day 28 to 35; LFU: Any day from Day 42 to Day 49
Population: Sepsis evaluable participants subset: participants who satisfied both clinical and microbiological criteria. Clinical: at least 1 criteria at Baseline, 1) body temperature >=38 or <36 degree Celsius, 2) WBC >12000 or <4000 cells/mm3, or immature neutrophil >10%, 3) heart rate >90 bpm, 4) SBP <90 mmHg, 5) CRP >=20 mg/dL. Microbiological: The most relevant pathogens isolated from blood at Baseline regardless of susceptibility.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06947386 + Metronidazole
Number analyzed (Participants) | 1
Participants
  EOT, Favorable | 1
  EOT, Unfavorable | 0
  EOT, Indeterminate | 0
  TOC, Favorable | 1
  TOC, Unfavorable | 0
  TOC, Indeterminate | 0
  LFU, Favorable | 1
  LFU, Unfavorable | 0
  LFU, Indeterminate | 0

35. Other Pre Specified Outcome: Percentage of Participants With Favorable Per-Pathogen Microbiological Response at EOT, TOC and LFU Visits: Sepsis Participants Subset
Description: Microbiological response: Favorable microbiological response assessments include "eradication", "presumed eradication" and "colonization". Unfavorable microbiological response assessments include "persistence", "persistence with increasing MIC", and "presumed persistence. Indeterminate: Study data was not available for evaluation of efficacy. EOT: within 24 hours after completion of last IV infusion. Response of baseline pathogens cultured from intra-abdominal site or blood. A participant can have more than 1 pathogen. LFU: after 42 calendar days from the day of the first IV infusion, the allowed visit window was 42 to 49 calendar days from the day of the first IV infusion. TOC: after 28 calendar days from the day of the first IV infusion, allowed visit window was 28 to 35 calendar days after the day of the first IV infusion.
Time Frame: EOT: 24 hours after last IV infusion; TOC: Any day from Day 28 to 35; LFU: Any day from Day 42 to Day 49
Population: Sepsis participants subset: participants who satisfied clinical & microbiological criteria; total score >=2 in SOFA for ICU participants, 2 items or more in qSOFA for non-ICU participants; most relevant pathogens (aerobic Gram-negative bacteria -either Enterobacterales or aerobic Gram-negative pathogens other than Enterobacterales) isolated from blood at Baseline regardless of susceptibility. "Number Analyzed": participants included in Sepsis participants subset at EOT & LFU respectively.
Measure: Number; unit: Percentage of Participants
Arm/Group | PF-06947386 + Metronidazole
Number analyzed (Participants) | 2
Percentage of Participants
  EOT, Escherichia Coli | 100.0
  EOT, Klebsiella Pneumoniae: number analyzed (Participants) | 1
  EOT, Klebsiella Pneumoniae | 100.0
  TOC, Escherichia Coli | 100.0
  TOC, Klebsiella Pneumoniae: number analyzed (Participants) | 1
  TOC, Klebsiella Pneumoniae | 100.0
  LFU, Escherichia Coli | 100.0
  LFU, Klebsiella Pneumoniae: number analyzed (Participants) | 1
  LFU, Klebsiella Pneumoniae | 100.0

36. Other Pre Specified Outcome: Number of Participants With Favorable Per-Pathogen Microbiological Response at EOT, TOC and LFU Visits: Sepsis Evaluation Participants Subset
Description: as for outcome 35
Time Frame: EOT: 24 hours after last IV infusion; TOC: Any day from Day 28 to 35; LFU: Any day from Day 42 to Day 49
Population: as for outcome 34
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06947386 + Metronidazole
Number analyzed (Participants) | 1
Participants
  EOT, Escherichia Coli | 1
  EOT, Klebsiella Pneumoniae | 1
  TOC, Escherichia Coli | 1
  TOC, Klebsiella Pneumoniae | 1
  LFU, Klebsiella Pneumoniae | 1
  LFU, Escherichia Coli | 1

37. Other Pre Specified Outcome: Number of Participants With Favorable Per-Pathogen Microbiological Response by MIC Categories at EOT, TOC and LFU Visits: Sepsis Participants Subset
Description: Microbiological response: Favorable microbiological response assessments include "eradication", "presumed eradication" and "colonization". Unfavorable microbiological response assessments include "persistence", "persistence with increasing MIC", and "presumed persistence. Indeterminate: Study data was not available for evaluation of efficacy. EOT: within 24 hours after completion of last IV infusion. LFU: after 42 calendar days from the day of the first IV infusion, the allowed visit window was 42 to 49 calendar days from the day of the first IV infusion. TOC: after 28 calendar days from the day of the first IV infusion, allowed visit window was 28 to 35 calendar days after the day of the first IV infusion.
Time Frame: EOT: 24 hours after last IV infusion; TOC: Any day from Day 28 to 35; LFU: Any day from Day 42 to Day 49
Population: Sepsis participants subset: participants who satisfied clinical & microbiological criteria: total score >=2 in SOFA for ICU participants, 2 items or more in qSOFA for non-ICU participants; most relevant pathogens isolated from blood at Baseline regardless of susceptibility. Here, "Number Analyzed" signifies participants included in Sepsis participants subset at EOT and LFU respectively.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06947386 + Metronidazole
Number analyzed (Participants) | 1
Participants
  EOT, Escherichia Coli, Susceptible | 1
  EOT, Escherichia Coli, Intermediate: number analyzed (Participants) | 0
  EOT, Escherichia Coli, Resistant: number analyzed (Participants) | 0
  EOT, Klebsiella Pneumoniae, Susceptible | 1
  EOT, Klebsiella Pneumoniae, Intermediate: number analyzed (Participants) | 0
  EOT, Klebsiella Pneumoniae, Resistant: number analyzed (Participants) | 0
  TOC, Escherichia Coli, Susceptible | 1
  TOC, Escherichia Coli, Intermediate: number analyzed (Participants) | 0
  TOC, Escherichia Coli, Resistant: number analyzed (Participants) | 0
  TOC, Klebsiella Pneumoniae, Susceptible | 1
  TOC, Klebsiella Pneumoniae, Intermediate: number analyzed (Participants) | 0
  TOC, Klebsiella Pneumoniae, Resistant: number analyzed (Participants) | 0
  LFU, Escherichia Coli, Susceptible | 1
  LFU, Escherichia Coli, Intermediate: number analyzed (Participants) | 0
  LFU, Escherichia Coli, Resistant: number analyzed (Participants) | 0
  LFU, Klebsiella Pneumoniae, Susceptible | 1
  LFU, Klebsiella Pneumoniae, Intermediate: number analyzed (Participants) | 0
  LFU, Klebsiella Pneumoniae, Resistant: number analyzed (Participants) | 0

38. Other Pre Specified Outcome: Number of Participants With Favorable Per-Pathogen Microbiological Response by MIC Categories at EOT, TOC and LFU Visits: Sepsis Evaluation Participants Subset
Description: as for outcome 37
Time Frame: EOT: 24 hours after last IV infusion; TOC: Any day from Day 28 to 35; LFU: Any day from Day 42 to Day 49
Population: as for outcome 34
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06947386 + Metronidazole
Number analyzed (Participants) | 1
Participants
  EOT, Klebsiella Pneumoniae, Susceptible | 1
  EOT, Klebsiella Pneumoniae, Intermediate: number analyzed (Participants) | 0
  EOT, Klebsiella Pneumoniae, Resistant: number analyzed (Participants) | 0
  TOC, Klebsiella Pneumoniae, Susceptible | 1
  TOC, Klebsiella Pneumoniae, Intermediate: number analyzed (Participants) | 0
  TOC, Klebsiella Pneumoniae, Resistant: number analyzed (Participants) | 0
  LFU, Klebsiella Pneumoniae, Susceptible | 1
  LFU, Klebsiella Pneumoniae, Intermediate: number analyzed (Participants) | 0
  LFU, Klebsiella Pneumoniae, Resistant: number analyzed (Participants) | 0

39. Other Pre Specified Outcome: Number of Participants With Treatment Emergent AEs and SAEs: Sepsis Participants Subset
Description: as for outcome 16
Time Frame: Up to Day 49
Population: as for outcome 33
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06947386 + Metronidazole
Number analyzed (Participants) | 2
Participants
  AEs | 2
  SAEs | 0

40. Other Pre Specified Outcome: Number of Participants With Treatment Emergent AEs and SAEs: Sepsis Evaluable Participants Subset
Description: as for outcome 16
Time Frame: Up to Day 49
Population: as for outcome 34
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06947386 + Metronidazole
Number analyzed (Participants) | 1
Participants
  AEs | 1
  SAEs | 0

ADVERSE EVENTS:
Time Frame: Up to Day 49
Description: Same event may appear as both an AE and SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another, or a participant may have experienced both a serious and non-serious event. Analysis performed on safety analysis set.
Arm/Group | PF-06947386 + Metronidazole
All-Cause Mortality (participants affected / at risk) | 1/60
Serious Adverse Events (participants affected / at risk) | 3/60
Other Adverse Events (participants affected / at risk) | 34/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-06947386 + Metronidazole (N=60)
Ileus (Gastrointestinal disorders) | 1
Pneumonia aspiration (Infections and infestations) | 1
Pyelonephritis (Infections and infestations) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Femur fracture (Injury, poisoning and procedural complications) | 1
Gout (Metabolism and nutrition disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PF-06947386 + Metronidazole (N=60)
Abdominal distension (Gastrointestinal disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 7
Diarrhoea (Gastrointestinal disorders) | 7
Nausea (Gastrointestinal disorders) | 4
Puncture site pain (General disorders) | 2
Pyrexia (General disorders) | 2
Incision site pain (Injury, poisoning and procedural complications) | 2
Wound complication (Injury, poisoning and procedural complications) | 4
Alanine aminotransferase increased (Investigations) | 2
Aspartate aminotransferase increased (Investigations) | 2
Blood magnesium abnormal (Investigations) | 2
Blood phosphorus abnormal (Investigations) | 2
Blood potassium abnormal (Investigations) | 2
Liver function test increased (Investigations) | 2
SARS-CoV-2 test positive (Investigations) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2
Headache (Nervous system disorders) | 2
Delirium (Psychiatric disorders) | 2
Insomnia (Psychiatric disorders) | 6
Blister (Skin and subcutaneous tissue disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 3
Hypertension (Vascular disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from the study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2021-07-21): https://cdn.clinicaltrials.gov/large-docs/12/NCT04927312/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-21): https://cdn.clinicaltrials.gov/large-docs/12/NCT04927312/SAP_001.pdf